CLINICAL TRIAL: NCT01491776
Title: Evaluation of the IND One Step Strep A Rapid Test Versus Culture Using Clinical Throat Swab Samples From Patients With Suspected Strep A Infections, CLIA Waiver Study
Brief Title: Evaluation of the IND One Step Strep A Rapid Test vs. Culture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IND Diagnostic Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IND-CSP-2011-01
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Strep Throat
Keywords: Group A Streptococcus; Strep A; Rapid Test; Pharyngitis
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to demonstrate the ability of the IND One Step Strep A test to accurately test a throat swab specimen from a symptomatic patient for the presence or absence of Group A Streptococcus (Strep A) when compared to culture.

DETAILED DESCRIPTION:
Group A Streptococcus is a principal cause of respiratory infections such as tonsillitis, pharyngitis, and scarlet fever. Since pharyngitis can lead to rheumatic fever or acute glomerulonephritis, it is important to differentiate streptococcal pharyngitis from viral disease during early stages of infection. The Strep A Rapid Test is a simple and rapid test which can detect Group A Streptococcal antigen directly from throat swabs allowing physicians to make a rapid diagnosis and to administer therapy immediately. The IND Diagnostic Inc. Strep A Rapid Test is a lateral flow immunoassay utilizing colloidal gold reagents labeled with Strep A antibody. The test detects either viable or nonviable organisms directly from throat swabs within 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects three (3) years of age or older
* Patients exhibiting at least 3 of the following symptoms:

  * fever
  * sore throat
  * swollen lymph nodes in the neck
  * redness of the throat and tonsils
  * white or yellow patches on the tonsils
* Must be able to collect 2 throat swab samples from patient

Exclusion Criteria:

* Patients currently undergoing antibiotic treatment will be excluded from study

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female subjects, 3 years of age or older, exhibiting symptoms consistent with Strep A infection.
Sampling Method: Non-Probability Sample
Enrollment: 315 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-03 (Estimated); Study Completion 2012-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Darin M. Gregory, MD, Principal Investigator — Pioneer Clinical Research; Sadia Dar, MD, Principal Investigator — HCCA Clinical Research; Sreedhar (Steve) Samudrala, MD, Principal Investigator — HCCA Clinical Research
Locations (3):
- United States (3):
  - Pioneer Clinical Research, LLC, Bellevue, Nebraska
  - HCCA Clinical Research, Franklin, Tennessee
  - HCCA Clinical Research, Smyrna, Tennessee